CLINICAL TRIAL: NCT03250910
Title: Generic Velpatasvir Plus Sofosbuvir With or Without Ribavirin for the Treatment of Hepatitis C Virus in Patients Coinfected With Human Immunodeficiency Virus
Brief Title: Generic VEL/SOF With or Without RBV for HIV/HCV Coinfected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201602026RINC
Record Dates: First submitted 2017-08-08; First posted 2017-08-16 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Hepatitis C Virus Infection, Response to Therapy of; Human Immunodeficiency Virus
Keywords: hepatitis C virus; human immunodeficiency virus; Direct acting antiviral agent
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome | interventions — sofosbuvir-velpatasvir drug combination; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HIV/HCV compensated liver disease (Experimental): Patients without cirrhosis or with compensated cirrhosis (Child-Pugh A) received a generic version of Sofosbuvir and Velpatasvir fixed-dose combination (Sofosvel®, VEL/SOF 100/400 mg film coated tablet, Beacon Pharmaceuticals Ltd. Mymensingh, Bangladesh) 1 tablet per day for 12 weeks.
  Interventions: Drug: Sofosbuvir and Velpatasvir
- HIV/HCV decompensated liver disease (Experimental): Patients with decompensated cirrhosis (Child-Pugh B or C) received Sofosvel® 1 tablet per day in combination with weight-based ribavirin (RBV)(Robatrol®, 200 mg capsule, Genovate Biotechnology Co. Ltd., Hsinchu, Taiwan; 1,200 mg per day if the body weight ≥ 75 kg; 1,000 mg per day if the body weight < 75 mg) for 12 weeks.
  Interventions: Drug: Sofosbuvir and Velpatasvir; Drug: Ribavirin
- HCV compensated liver disease (Active Comparator): Patients without cirrhosis or with compensated cirrhosis (Child-Pugh A) received a generic version of Sofosbuvir and Velpatasvir fixed-dose combination (Sofosvel®, VEL/SOF 100/400 mg film coated tablet, Beacon Pharmaceuticals Ltd. Mymensingh, Bangladesh) 1 tablet per day for 12 weeks.
  Interventions: Drug: Sofosbuvir and Velpatasvir
- HCV decompensated liver disease (Active Comparator): Patients with decompensated cirrhosis (Child-Pugh B or C) received Sofosvel® 1 tablet per day in combination with weight-based ribavirin (RBV)(Robatrol®, 200 mg capsule, Genovate Biotechnology Co. Ltd., Hsinchu, Taiwan; 1,200 mg per day if the body weight ≥ 75 kg; 1,000 mg per day if the body weight < 75 mg) for 12 weeks.
  Interventions: Drug: Sofosbuvir and Velpatasvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir and Velpatasvir — All patients received a generic version of VEL/SOF fixed-dose combination (Sofosvel®, VEL/SOF 100/400 mg film coated tablet, Beacon Pharmaceuticals Ltd. Mymensingh, Bangladesh) 1 tablet per day for 12 weeks.
  Other Names: Sofosvel
Drug: Ribavirin — Patients with decompensated cirrhosis (Child-Pugh B or C), received weight-based ribavirin (RBV)(Robatrol®, 200 mg capsule, Genovate Biotechnology Co. Ltd., Hsinchu, Taiwan; 1,200 mg per day if the body weight ≥ 75 kg; 1,000 mg per day if the body weight < 75 mg) for 12 weeks.
  Other Names: Robatrol
  Arms: HCV decompensated liver disease; HIV/HCV decompensated liver disease

SUMMARY:
Data are limited regarding the effectiveness and safety of generic velpatasvir plus sofosbuvir (VEL/SOF) with or without ribavirin (RBV) for the treatment of hepatitis C virus (HCV) in patients with human immunodeficiency virus (HIV) coinfection. We aim to compare the effectiveness and safety of VEL/SOF with and without RBV for 12 weeks in HIV/HCV-coinfected and HCV-monoinfected patients The antiviral responses and the adverse events (AEs) are compare between the two groups. The characteristics potentially related to sustained virologic response 12 weeks off therapy (SVR12) are analyzed.

DETAILED DESCRIPTION:
Due to the lack of effective vaccination and the shared routes of transmission, hepatitis C virus (HCV) infection remains a challenging co-morbidity in patients with human immunodeficiency virus (HIV) infection. It is estimated that approximately 2.3 million people are coinfected with HIV and HCV (HIV/HCV) in the world. Compared to patients with HCV monoinfection, HIV/HCV-coinfected patients tend to have higher serum HCV viral loads, faster hepatic fibrosis progression, and higher risks of hepatic decompensation. Following the commencement of scale-up antiretroviral therapy (ART) that decreases the HIV-related opportunistic infections and malignancies, the liver-related complications have now become the leading cause of morbidity and mortality in HIV/HCV-coinfected patients. On the other hand, the survival rate is improved if these patients achieve sustained virologic response (SVR) by anti-HCV agents.

On the basis of excellent efficacy and safety, treatment by interferon (IFN)-free direct acting antiviral agents (DAAs) has made a paradigm shift for HCV care. Velpatasvir (VEL) is an HCV non-structural protein 5A (NS5A) inhibitor and sofosbuvir (SOF) is an HCV NS5B nucleotide polymerase inhibitor. Both agents are active against HCV with pan-genotypic potency. A fixed-dose combination of VEL at a daily dosage of 100 mg and SOF at a daily dosage of 400 mg (VEL/SOF) with or without weight-based ribavirin (RBV) has been approved by U.S. Food and Drug Administration (FDA) and European Medicines Agency (EMA) to treat HCV genotype 1-6 patients with compensated and decompensated liver diseases, respectively. Recently, a phase 3 study of VEL/SOF to treat HCV infection in HIV-coinfected patients reveals that this regimen is safe and provides a high and comparable SVR rate to HCV-monoinfected patients.

Although treatment of HCV by IFN-free DAAs is considered highly efficacious and well tolerated, numerous HCV-infected individuals have limited access to the brand-name agents due to the lack of universal governmental reimbursement or private insurance support. Therefore, allowing the generic version of patented DAAs for HCV through voluntary or compulsory licensing may provide patients with greater access to new HCV treatment, particularly in resource-constrained countries. Regarding the real-world experiences of generic IFN-free DAAs, a recent report from China evaluated the effectiveness of a generic version of ledipasvir (LDV) plus SOF (LDV/SOF) with or without RBV for 8-12 weeks in 192 HCV genotype 1b (HCV-1b) patients. The overall SVR rates were excellent (96.8%-96.9%) and most patients tolerated the treatment well. Based on the encouraging results, we aim to evaluate the effectiveness and safety of a generic version of pan-genotypic VEL/SOF-based therapy for HCV in HIV-coinfected patients, and compare the performance of such a regimen in HCV-monoinfected patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 20 years
* Chronic HCV infection, defined as detectable HCV antibody (anti-HCV; Abbott HCV EIA 2.0, Abbott Laboratories, Abbott Park, Illinois, USA) and quantifiable serum HCV RNA (Cobas TaqMan HCV Test v2.0, Roche Diagnostics GmbH, Mannheim, Germany, lower limit of quantification [LLOQ]: 25 IU/mL) for ≥ 6 months

Exclusion Criteria:

* Chronic kidney disease (CKD) stage ≥ 4,
* Organ transplantation
* Prior DAA exposure
* Refusal to provide written informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response | 24 weeks
  HCV RNA < LLOQ 12 weeks off therapy

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Hua Liu, MD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Yun-Lin Branch, Douliu
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No